CLINICAL TRIAL: NCT06520735
Title: Effect of Transcutaneous Electrical Nerve Stimulation Versus Capsicum Plaster on Emesis Gravidarum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Peter Bahgat Milad, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003610
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2024-08

CONDITIONS: Emesis Pregnancy
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous electrical nerve stimulation group (Experimental): The pregnant women with emesis gravidarum will be treated by transcutaneous electrical nerve stimulation on the P6 acupuncture point.
  Interventions: Device: Transcutaneous electrical nerve stimulation
- Capsicum plaster group (Experimental): The pregnant women with emesis gravidarum will be treated with capsicum plaster on the P6 acupuncture point.
  Interventions: Other: Capsicum plaster

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — The pregnant women with emesis gravidarum will be treated by transcutaneous electrical nerve stimulation (TENS) on p6 acupuncture point for 30 minutes daily for 5 consecutive days.
  Arms: Transcutaneous electrical nerve stimulation group
Other: Capsicum plaster — The pregnant women with emesis gravidarum will be treated with capsicum plaster on p6 acupuncture point for 12 hours per day for 5 consecutive days.
  Arms: Capsicum plaster group

SUMMARY:
This study will be conducted to determine the difference between the effect of transcutaneous electrical nerve stimulation and capsicum plaster on emesis gravidarum.

DETAILED DESCRIPTION:
Almost 50-90% of pregnant women experience nausea vomiting in the first trimester. Nausea vomiting occurs in 60% -80% primigravida and 40% -60% in multigravida.It is revealed that 50% of affected women have a significant reduction of their work efficiency.

Transcutaneous acupoint electrical stimulation (TAES) at the Nei-Guan P6 acupoint may be a useful alternative to antiemetic drugs. It is effective in the treatment of both motion sickness and pregnancy induced nausea and vomiting , as well as emesis associated with chemotherapy.

Capsicum plaster is an alternative to acupuncture. It is applied to the acupuncture points and has been reported to be an effective method for preventing postoperative nausea and vomiting (PONV), postoperative sore throat, and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women complaining of emesis gravidarum
* Their ages will be ranged from 20 to 35 years old.
* Their body mass index will not exceed 35 kg/ m2.
* Their gestational age will be less than 20 weeks.
* All women having mild to moderate nausea and/or vomiting
* All women having singleton pregnancy

Exclusion Criteria:

Women will be excluded from the study if they have:

* Previous carpal tunnel syndrome.
* Skin abnormalities
* Acute viral disease
* Hyperemesis gravidarum.
* Previous history of nausea or vomiting before pregnancy.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Rhodes index for nausea and vomiting and retching | within Five days
  It will be used to assess the severity of nausea (N), vomiting (V) and retching (R) for both groups before and after treatment.
  It is an instrument consisting of eight 5-point self report items measuring the individual's perception of duration of nausea, frequency of nausea, distress from nausea, frequency of vomiting, amount of vomiting, distress from vomiting, frequency of retching, and distress from retching.
  Its score ranges from 0 to 32. A score of 0 indicated no nausea, vomiting, or retching (NVR), 1-8 indicated mild NVR, 9-16 indicated moderate NVR, 17-24 indicated severe NVR, and 24-32 indicated the worst levels of NVR.
Modified pregnancy unique quantification of emesis and nausea (MPUQE) | within five days
  Nausea and vomiting of pregnancy (NVP) were measured and classified into three groups of different severity by using the 24-h Modified Pregnancy Unique Quantification of Emesis Scale (PUQE). MPUQE consists of three items that are used to assess the severity of NVP; the number of hours of nausea, the number of episodes of retching, and the number of episodes of vomiting within the last 24 hours. Each item has five options which are scored from 1 to 5 points. The MPUQE score is calculated by adding the values from each item which adds up to a total score that ranges from 3 to 15 points. The obtained total MPUQE-score was used to classify the severity of NVP into mild ≤6 points; moderate 7-12 points; severe ≥13 points.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Emara, professor, Study Chair — Cairo University; Mohamed Awad, professor, Study Director — Cairo University; Amir Arabi, professor, Study Director — Cairo University
Locations (1):
- Peter Bahgat Milad, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol